CLINICAL TRIAL: NCT06545825
Title: Effects of Prolonged and Chronic Critical Illness Induced by Brain Injury on Metabolic State: Matched Case-control Study
Brief Title: Effects of Prolonged and Chronic Critical Illness Induced by Brain Injury on Metabolic State
Status: Completed | Type: Observational
Sponsor: Federal Research and Clinical Centre of Intensive Care Medicine and Rehabilitology (Other)
Responsible Party: Sponsor
Other Study IDs: PRIME-Met
Record Dates: First submitted 2024-08-06; First posted 2024-08-09 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Brain Injuries; Stroke; Malnutrition; Critical Illness
Keywords: Brain Injuries; Stroke; Malnutrition; Prolonged critical illness; Chronic critical illness
MeSH Terms: conditions — Brain Injuries; Stroke; Malnutrition; Critical Illness

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Standard enteral nutrition: Patients with prolonged or chronic critical illness and brain injury receiving standard enteral nutrition
  Interventions: Other: Standard enteral nutrition

INTERVENTIONS:
Other: Standard enteral nutrition — Enteral nutrition will be given with standard isocaloric mixtures. Mixture volume calculation will be performed after indirect calorimetry, adjusted for daily nitrogen loss.

SUMMARY:
Brain injuries, including acute stroke (AS) and traumatic brain injury (TBI), are prevalent pathologies with severe consequences. Cerebral infarction accounts for 65-85% of AS cases, while hemorrhagic stroke, though less common, has a higher mortality rate (30-50%) and limited recovery (10-20%). TBI is a significant medical and socioeconomic issue due to its high prevalence, severe consequences, and the high rates of temporary and permanent disability, particularly among young and working-age adults. The average mortality rate for severe TBI is 39%, with 60% facing unfavorable outcomes according to the Glasgow Outcome Scale.

High levels of permanent disability, a low percentage of patients returning to work, and long-term rehabilitation after brain injury impose a heavy economic and social burden. Severe brain damage often leads to chronic critical illness (CCI), a term introduced in 1985 to describe patients with prolonged ICU stays. CCI affects 6-10% of ICU patients, with an increasing prevalence. About 5-10% of those requiring mechanical ventilation develop CCI, with a significant number following sepsis. The prevalence of CCI is estimated at 34.4 to 42.0 cases per 100,000 people, increasing with age.

Malnutrition and the hypermetabolism-hypercatabolism syndrome are major complications in AS and TBI, leading to poor treatment outcomes and extended recovery periods. Effective rehabilitation is impossible without adequate nutritional support. Despite the universal metabolic response to different types of damage, specific metabolic disorders vary among different pathological conditions, both in macro- and micronutrient exchange.

Developing specialized enteral nutrition products tailored to specific conditions, like brain injury, is of great scientific and practical interest. To advance this development, comprehensive data on metabolic disorders in these patients is essential.

DETAILED DESCRIPTION:
Brain injury is a common pathology and is most often represented by acute stroke (AS) and traumatic brain injury (TBI). 65-85% of diagnosed acute stroke is cerebral infarction. Hemorrhagic stroke is less common, but its mortality is higher. Mortality in hemorrhagic stroke ranges from 30 to 50%, and recovery of functional activity is only in 10-20%. TBI remains a serious medical and socioeconomic problem because of prevalence and severity of consequences, high levels of temporary and permanent disability, and high mortality rates. TBI is the most common death reason and disability among young and adult people, as it is the most active part of the population in work and social relations. The average weighted mortality rate for severe TBI is 39%, and for an unfavorable outcome according to the Glasgow Outcome Scale (GOS) - 60%. TBI ranks first in mortality and disability among the population under 44 years of age.

The high level of permanent disability, low percentage of patients returning to work, long-term rehabilitation after brain injury is a heavy economic and social burden. Severe brain damage can also lead to the development of prolonged/chronic critical illness.

In 1985, scientists first described the characteristics of patients who spent a long time in the intensive care unit (ICU) and introduced the term "chronically critically ill". Then many authors introduced the terms prolonged critical illness, protracted critical illness, which meant a long-term or prolonged critical condition. Of the total number of ICU patients, 6 to 10% are patients with chronic critical illness syndrome (CCI). It should be noted that the proportion of this category of patients in ICUs has tended to increase in recent years. It is estimated that 5-10% of patients who require mechanical ventilation as part of their initial illness will go on to develop prolonged/CCI. More than a third of patients after sepsis, and in particular after abdominal sepsis, develop prolonged/CCI, and according to Canadian authors, this condition develops in one in six intensive care patients. The overall prevalence is estimated at 34.4 cases per 100,000 population, and according to Japanese authors it reaches 42.0 cases per 100,000 population (this figure steadily increases with age, reaching 109.6 cases per 100,000 population over 85 years of age).

Malnutrition and metabolic response to stress as the form of hypermetabolism-hypercatabolism syndrome are among the leading complications and one of the main links in AS's and TBI's pathogenesis. These determine the unfavorable course and results of treatment of this category of patients. In this time that syndrome is considered both as an independent cause of death and as a factor provoking a large number of complications. Malnutrition significantly extends the treatment period and also affects the recovery process. So it's impossible to perform effective rehabilitation without nutritional support.

Although the metabolic response is universal to different types of damage, many studies indicate that there are certain features of metabolic disorders in different pathological conditions. This is true for both macro- and micronutrient exchange. Therefore, the development of specialized enteral nutrition products with a metabolic focus on a specific pathological condition, in particular brain injury, is of great scientific and practical interest.

Thus, in order to move on to the development of such products, it is necessary to obtain data on the full picture of metabolic disorders in this category of patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient's age is between 18 and 74
* Stay in the intensive care unit >5 days from the time of injury
* Presence of brain injury or stroke
* Receiving enteral nutrition
* Informed voluntary consent of the patient to participate in the study, or a decision of the medical council to include the patient in the study

Exclusion Criteria:

* Diabetes mellitus
* Acute kidney injury
* Acute liver failure
* Shock of any etiology
* Presence of a cardiac implantable electronic device or neurostimulator
* Presence of a tracheoesophageal fistula
* Positive end expiratory pressure > 12 mbar
* Patients previously included in this trial

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with prolonged or chronic critical illness and brain injury receiving standard enteral nutrition
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2024-09-09 (Actual); Primary Completion 2024-10-24 (Actual); Study Completion 2024-11-15 (Actual)

PRIMARY OUTCOMES:
Change from baseline in serum level of total protein | From day 1 to day 20
  The serum level of total protein is measured in g/L. Normal values range from 65 to 85 g/L.

SECONDARY OUTCOMES:
Change from baseline in serum level of albumin | From day 1 to day 20
  The serum level of albumin is measured in g/L. Normal values range from 35 to 52 g/L
Change from baseline in serum level of transferrin | From day 1 to day 20
  The serum level of transferrin is measured in g/L. Normal values range from 2.0 to 3.6 g/L
Change from baseline in serum level of glucose | From day 1 to day 20
  The serum level of glucose is measured in mmol/L. Normal values range from 3.3 to 6.5 mmol/L
Change from baseline in serum level of cholesterol | From day 1 to day 20
  The serum level of cholesterol is measured in mmol/L. Normal values are less than 5.2 mmol/L
Change from baseline in serum level of very low density lipoprotein | From day 1 to day 20
  The serum level of very low density lipoprotein is measured in mg/dL. Normal values range from 2 to 30 mg/dL
Change from baseline in serum level of low density lipoprotein | From day 1 to day 20
  The serum level of low density lipoprotein is measured in mg/dL. Normal values are less than 100 mg/dL
Change from baseline in serum level of high density lipoprotein | From day 1 to day 20
  The serum level of high density lipoprotein is measured in mg/dL. Normal values are greater than 60 mg/dL.
Change from baseline in absolute lymphocyte count | From day 1 to day 20
  absolute lymphocyte count is measured in lymphocytes per microliter. Normal values range from 1,000 to 4,800 lymphocytes per microliter.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Shestopalov, PhD, Principal Investigator — Federal Research and Clinical Centre of Intensive Care Medicine and Rehabilitology
Locations (1):
- Federal Research and Clinical Centre of Intensive Care Medicine and Rehabilitology, Moscow, Moscow Oblast, Russia

IPD SHARING:
Plan to Share IPD: No